CLINICAL TRIAL: NCT06516744
Title: A Single Group Study to Evaluate the Efficacy of Bye Bye Bloat Capsules in Relieving Bloating and Promoting Healthy Digestion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Love Wellness (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20402
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Digestive Health; Digestion
Keywords: Gastrointestinal Symptoms; Hormonal Bloating; Capsule Supplement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bye Bye Bloat Capsules (Experimental): Participants will take 2 Bye Bye Bloat capsules immediately after eating (when they feel full and bloated) at least 3 times a week. They may also take the product during times of hormonal bloating. The study will last for 4 weeks, with questionnaires and waist measurements completed at Baseline, first use, Week 2, and Week 4.
  Interventions: Dietary Supplement: Bye Bye Bloat Capsules

INTERVENTIONS:
Dietary Supplement: Bye Bye Bloat Capsules — Bye Bye Bloat Capsules contain the following ingredients: Organic Fenugreek Seed Powder, Organic Dandelion Root Powder, Organic Fennel Seed Powder, Organic Ginger Root Powder, Organic Parsley Leaf Powder, Amylase Complex, Protease Complex, Pepsin Complex, Lipase Complex, Bromelain Complex, Papain Complex. Other ingredients include Hypromellose Capsule, Maltodextrin, Microcrystalline Cellulose, and Magnesium Stearate. Participants will take 2 capsules immediately after eating at least 3 times a week and during times of hormonal bloating for 4 weeks.

SUMMARY:
This virtual single-group study aims to evaluate the efficacy of Bye Bye Bloat Capsules in relieving hormonal and food-related bloating and promoting healthy digestion. The study will last 4 weeks, involving 40 female participants aged 18+ who will take two capsules after meals and during times of bloating. Measurements and questionnaires will be completed at Baseline, first use, Week 2, and Week 4.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18+
* Self-reported concerns with bloating after eating
* Issues with hormonal bloating
* Generally healthy without uncontrolled chronic diseases
* Willing to avoid using digestive health remedies and other oral supplements during the study

Exclusion Criteria:

* Pre-existing chronic conditions preventing adherence to the protocol
* Undergoing procedures related to digestive health
* Started new medications or supplements targeting digestive health in the past 3 months
* Severe allergic reactions requiring an Epi-Pen
* Pregnant, breastfeeding, or attempting to conceive
* Unwilling to follow the study protocol
* Recent surgeries or planned surgeries during the study
* Diagnosed gastrointestinal disorders
* Recent changes in hormonal birth control use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Reduction in Bloating | Baseline, first use, Week 2, and Week 4
  Evaluation of parameters associated with hormonal and food-related bloating through self-reported questionnaires taken at Baseline, first use, Week 2, and Week 4.

SECONDARY OUTCOMES:
Improvement in Digestion and Mental Well-being | Baseline, first use, Week 2, and Week 4
  Assessment of changes in participant perception of digestion, gas, mental health, and well-being associated with bloating through self-reported questionnaires taken at Baseline, first use, Week 2, and Week 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No